CLINICAL TRIAL: NCT01006798
Title: Phase 1 Evaluation of the Safety and Immunogenicity of a Replication-Competent Adenovirus Serotype 4-vectored H5N1 Influenza Candidate Vaccine - Ad4-H5-Vtn
Brief Title: Safety and Immunogenicity of Replication-Competent Adenovirus 4-vectored Vaccine for Avian Influenza H5N1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PXVX-H5-103-001
Record Dates: First submitted 2009-11-02; First posted 2009-11-03 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Bird Flu; Influenza
Keywords: Virus Diseases; Respiratory Tract Diseases; Vaccine
MeSH Terms: conditions — Influenza in Birds; Influenza, Human; Virus Diseases; Respiratory Tract Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1 (Experimental): three vaccinations of 10^7vp Ad4-H5-Vtn or placebo
  Interventions: Other: Placebo; Biological: Ad4-H5-Vtn; Biological: Sanofi Pasteur Influenza Virus Vaccine, H5N1
- Cohort 2 (Experimental): three vaccinations of the 10^8vp Ad4-H5-Vtn or placebo
  Interventions: Other: Placebo; Biological: Ad4-H5-Vtn; Biological: Sanofi Pasteur Influenza Virus Vaccine, H5N1
- Cohort 3 (Experimental): three vaccinations of 10^9 Ad4-H5-Vtn or placebo
  Interventions: Other: Placebo; Biological: Ad4-H5-Vtn; Biological: Sanofi Pasteur Influenza Virus Vaccine, H5N1
- Cohort 4 (Experimental): three vaccinations of 10^10 Ad4-H5-Vtn or placebo
  Interventions: Other: Placebo; Biological: Ad4-H5-Vtn; Biological: Sanofi Pasteur Influenza Virus Vaccine, H5N1
- Cohort 5 (Experimental): three vaccinations of 10^11 Ad4-H5-Vtn or placebo
  Interventions: Other: Placebo; Biological: Ad4-H5-Vtn; Biological: Sanofi Pasteur Influenza Virus Vaccine, H5N1

INTERVENTIONS:
Other: Placebo — enteric coated capsule containing no vaccine virus
  Other Names: Placebo for Ad4-H5-Vtn
Biological: Ad4-H5-Vtn — a live, replication-competent, recombinant Ad4 virus expressing the HA of H5N1 influenza (A/Vietnam/1194/2004) in an enteric capsule for oral administration
  Other Names: Adenovirus Serotype 4-vectored H5N1 Influenza Vaccine
Biological: Sanofi Pasteur Influenza Virus Vaccine, H5N1 — Single administration of a heterologous boost given to volunteers 3 to 15 months following their last vaccination with Ad4-H5-Vtn or placebo.
  Other Names: FDA-licensed inactivated monovalent Influenza Virus Vaccine, H5N1; licensed H5N1 vaccine

SUMMARY:
The purpose of this study is to compare the safety and immunogenicity over a 9-month period of five different dosages of Ad4-H5-Vtn in volunteers (Vaccinees) who receive three doses of the study vaccine or placebo. In addition, transmission of Ad4-H5-Vtn will be evaluated in all Household Contacts residing with the vaccinated volunteers.

Vaccinees also may participate in a substudy in which they receive a booster vaccination with the licensed Influenza Virus Vaccine, H5N1 (Sanofi Pasteur).

DETAILED DESCRIPTION:
At least 160 healthy Vaccinees will be randomized into 5 ascending dosage cohorts each consisting of at least 32 volunteers. In each dosage cohort Vaccinees will be randomly assigned to receive 3 doses of either Ad4-H5-Vtn or placebo separated by approximately 56 days. Volunteers will be followed for 168 days post-third vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults and their healthy adult household contacts.

Exclusion Criteria:

* Healthcare workers who have direct contact with patients who are immunodeficient, are HIV-positive, have an unstable medical condition, or are under the age of 18.
* Childcare workers who have direct contact with children 5 years old and younger.
* Resides with Household Contacts who are under the age of 18 or over the age of 65.
* Received or plans to receive licensed inactivated 2009 H1N1 influenza vaccine from 14 days prior to 14 days after any study vaccination.
* Received or plans to receive any other licensed vaccines from 30 days prior to the first study vaccination until 30 days after the third study vaccination.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 166 (Actual)
Dates: Start 2009-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Safety, defined as the frequency and severity of vaccine-related reactogenicity events and reported AEs | Throughout trial (reactogenicity for 7 days following each vaccination)
Immunogenicity (humoral) defined by H5 HAI titer | At all available timepoints

SECONDARY OUTCOMES:
Immunogenicity (humoral), defined by Ad4 antibody response | At all available timepoints
Replication/excretion of Ad4-H5-Vtn virus | Throughout trial
Transmission to household contacts as measured by AE assessment and antibody response and viral replication/excretion | Throughout trial

CONTACTS AND LOCATIONS:
Overall Officials: Marc Gurwith, M.D., J.D., Study Director — Emergent BioSolutions
Locations (4):
- United States (4):
  - University of Kentucky, Lexington, Kentucky
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - University of Rochester, Rochester, New York
  - Coastal Carolina Research Center, Inc., Mt. Pleasant, South Carolina

REFERENCES:
- [Background] Khurana S, Coyle EM, Manischewitz J, King LR, Ishioka G, Alexander J, Smith J, Gurwith M, Golding H. Oral priming with replicating adenovirus serotype 4 followed by subunit H5N1 vaccine boost promotes antibody affinity maturation and expands H5N1 cross-clade neutralization. PLoS One. 2015 Jan 28;10(1):e0115476. doi: 10.1371/journal.pone.0115476. eCollection 2015. PMID 25629161
- [Result] Gurwith M, Lock M, Taylor EM, Ishioka G, Alexander J, Mayall T, Ervin JE, Greenberg RN, Strout C, Treanor JJ, Webby R, Wright PF. Safety and immunogenicity of an oral, replicating adenovirus serotype 4 vector vaccine for H5N1 influenza: a randomised, double-blind, placebo-controlled, phase 1 study. Lancet Infect Dis. 2013 Mar;13(3):238-50. doi: 10.1016/S1473-3099(12)70345-6. Epub 2013 Jan 29. PMID 23369412